CLINICAL TRIAL: NCT07026942
Title: A Phase I/II Clinical Trial Evaluating the Safety and Efficacy of Universal Donor CD33 CAR Natural Killer Cells for Treatment of Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Phase I/II Clinical Trial of Universal Donor CD33 CAR Natural Killer Cells for AML
Acronym: CD33 CAR NK
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Margaret Lamb, Assistant Professor of Pediatrics, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD33 CAR NK
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Relapsed/Refractory AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: A single-arm, unblinded, dose escalation study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CD33 CAR NK Cells (Experimental): Patients will undergo 5 days of lymphodepleting chemotherapy (Fludarabine and Cytarabine) along with oral Venetoclax given from days 1-21 of the cycle.
  CD33 CAR NK cells will be infused on day 7 (and day 14 for dose level 4).
  Dose Levels
  * Dose level 1: 1 x 10^7 CD33 CAR-NK cells/kg
  * Dose level 2: 3 x 10^7 CD33 CAR-NK cells/kg
  * Dose level 3: 1 x 10^8 CD33 CAR-NK cells/kg
  * Dose level 4: 2 doses of 1 x 10^8 CD33 CAR-NK cells/kg
  Interventions: Biological: Universal donor derived CD33 CAR-NK

INTERVENTIONS:
Biological: Universal donor derived CD33 CAR-NK — Universal donor derived CD38KO CD33 CAR-NK manuctured on-site. The NK cells are derived from the peripheral blood of universal donors with desirable HLA/KIR types and CMV status, modified by CRISPR/Cas9 targeting the CD38 locus, using AAV6 vector to insert a CD33-targeted CAR gene into the CD38 locus, and expanded in number.

SUMMARY:
This phase 1/2 study is testing a new treatment for acute myeloid leukemia (AML) that has come back or has not responded to other treatments. The treatment uses specially modified immune cells (called CD33 CAR-NK cells) from a healthy, unrelated donor to attack the cancer.

The first part of the study (Phase I) will focus on finding the safest and most effective dose. The second part (Phase II) will test how well the treatment works at that dose.

Patients will undergo screening, chemotherapy (Fludarabine and Cytarabine, in combination with Venetoclax) followed by the infusion of the CD33 CAR NK cells. Some patients may receive 2 doses of CD33 CAR NK cells infused 1 week apart. The investigator will let participants know if they will receive 1 or 2 doses. Patients will be hospitalized for the chemotherapy and CD33 CAR NK cell infusion for close monitoring and will remain in the hospital until blood counts recover. If patients are discharged from the hospital before day 35, they will be followed in clinic weekly for blood work and a physical exam.

A bone marrow biopsy will be performed around day 28-35 to see if the patient's leukemia is in remission. Lumbar puncture or imaging may also be done if the study doctor thinks it is necessary.

Patients will continue to be followed for research studies and clinical outcomes (leukemia relapse, survival) for 1 year. After 1 year, patients will have completed their study participation, but can be monitored for up to 15 years for potential long term side effects of the cell therapy. Some patients may undergo a bone marrow transplant after the study treatment. Patients who proceed to bone marrow transplant will have one blood sample drawn about a month after the transplant and then will have completed study participation.

DETAILED DESCRIPTION:
This is a phase I/II study designed to determine the safety and estimate the efficacy of CD33 CAR-NK cells combined with FLA-VEN chemotherapy in patients age 1-39.99 with relapsed or refractory acute myeloid leukemia. This study will be performed in two phases: a dose-finding phase and a phase II expansion phase to further study safety and estimate efficacy. To determine the recommended phase II dose investigators will utilize a Bayesian optimal interval (BOIN) dose escalation design. Once a RP2D is established, a phase II expansion cohort of 24 total patients will be enrolled to evaluate efficacy and correlative data while also continually gathering data on safety and toxicity.

Manufacturing of the CD33 CAR NK Cells:

NK cells are derived from the peripheral blood of universal donors with desirable HLA/KIR types and CMV status, modified by CRISPR/Cas9 targeting the CD38 locus, using AAV6 vector to insert a CD33-targeted CAR gene into the CD38 locus, and expanded in number.

Dose Levels

* Dose level 1: 1 x 10^7 CD33 CAR-NK cells/kg
* Dose level 2: 3 x 10^7 CD33 CAR-NK cells/kg
* Dose level 3: 1 x 10^8 CD33 CAR-NK cells/kg
* Dose level 4: 2 doses of 1 x 10^8 CD33 CAR-NK cells/kg

Chemotherapy:

Days 1-5: Fludarabine 30 mg/m2/d, cytarabine 2g/m2/d Days 1-21: Venetoclax Day 7: CD33 CAR NK infusion Day 14; CD33 CAR NK infusion (for patients on DL4)

Patients will be admitted to the hospital for 4-5 weeks during each cycle of treatment for count nadir and recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with relapsed or primary refractory CD33+ AML, including:

   * Patients with relapsed AML (patients in second or subsequent relapse, or any relapse after HSCT, are eligible).
   * Refractory AML defined as failure to achieve a complete response after 2 cycles of induction or reinduction chemotherapy, including persistent MRD positivity.
   * Patients with isolated CNS or extramedullary disease are eligible. Patients with CNS disease are excluded from the phase I dose escalation portion but are eligible for the phase II portion of the study.
2. 1-39.99 years of age (note: the first three subjects treated AND the first subject on each dose level must be ≥ 16 years of age)
3. Negative serum test to rule out pregnancy within 14 days prior to enrollment in females of childbearing potential

   o Sexually active males and females of childbearing potential must agree to use a form of contraception considered effective and medically acceptable by the Investigator for 6 months after the last dose of chemotherapy and/or NK cell infusion
4. Organ function requirements:

   * Renal function: Creatinine ≤ 2 times the institutional upper limit of normal for age OR creatinine clearance > 60 ml/min/1.73m2 (measured by 24 hour- urine specimen or radioisotope GFR)
   * Liver function: Total bilirubin ≤ 2 mg/dl (unless Gilbert's syndrome), AST and ALT ≤ 5 times the upper limit of normal (unless related to leukemic involvement). Upper limit of normal should be determined by the institutional defined normal laboratory range.
   * Cardiac function: left ventricular ejection fraction ≥ 40% or shortening fraction ≥20%. May be eligible after cardiology clearance if qualitatively normal function or repeat measures are normal.
   * CNS: Patients with seizure disorder may be eligible if seizures are well controlled
   * Pulmonary function: baseline oxygen saturation >92% on room air at rest
5. Due to the risk of hematopoietic toxicity from CD33 targeting, enrolled subjects must have an allogeneic HCT donor identified and be eligible and willing to undergo a subsequent HSCT in the event of aplasia.
6. All patients or their legal guardian must be able to understand and willing to sign a written informed consent document.
7. All patients must consent to enroll in a separate long term follow up study for cell and gene therapy

Exclusion Criteria:

1. Prior therapies:

   * AML directed therapies in the 14 days prior to beginning treatment on this protocol (except for hydroxyurea) Note: There is no waiting period required for patients having received intrathecal cytarabine, methotrexate and/or hydrocortisone
   * Gemtuzumab or other CD33-targeted antibody within 42 days of enrollment
   * CNS radiation within 28 days of enrollment
   * DLI or adoptive cell therapy within 30 days of enrollment
   * Allogeneic SCT within 90 days of enrollment

     * Patients with CNS disease are excluded from the phase I portion of the study but are eligible for the phase II expansion phase.
     * Patients on immunosuppressive therapy
   * Patients must be off of systemic immunosuppressive therapy for at least 14 days prior to enrollment with no evidence of recurrent GVHD
   * Patients on hydrocortisone for treatment of adrenal insufficiency are permitted on study
   * Patients on corticosteroids ≤ 0.5mg/kg/day (prednisone equivalent) for any other indication are permitted on study
2. Uncontrolled, symptomatic, intercurrent illness or social situations that would limit compliance with study requirements or in the opinion of the site PI would pose an unacceptable risk to the subject
3. Patients who are breastfeeding
4. Patients with prior solid organ transplantation
5. Performance status: Karnofsky or Lansky Performance Scale (PS) < 50
6. Uncontrolled infection, defined as an infection which has not resolved or does not show evidence of significant resolution after initiating appropriate therapy

   o Asymptomatic viremia such as CMV, HPV, BK virus, HCV, etc. is NOT considered as an exclusion criterion
7. Uncontrolled arrhythmias or uncontrolled symptomatic cardiac disease
8. Active acute or chronic GVHD of any grade at the time of enrollment. "Active GVHD" is defined as a patient who requires immunosuppressive therapy for control of their GVHD symptoms.

Ages: 1 Year to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2032-07-01 (Estimated); Study Completion 2038-07-01 (Estimated)

PRIMARY OUTCOMES:
Phase I : Safety and recommended phase 2 dose | From the first CD33 CAR NK cell infusion until 28 days after the last CAR NK cell dose.
  To determine the safety and recommended phase 2 dose of CD33 CAR-NK cells in patients with relapsed/refractory AML investigators will monitor the incidence and severity of adverse events and the rate of dose limiting toxicities.
Phase II: Efficacy of CD33 CAR NK cells | Day 35
  To estimate the efficacy of CD33 CAR-NK cells delivered at the RP2D with FLA-VEN chemotherapy, the investigators will determine the complete response rate.

SECONDARY OUTCOMES:
Overall survival, event free survival and duration of remission | 1 year
  To estimate the overall survival, event free survival, and duration of remission in patients who do not proceed to HSCT.
Depth of remission | Day 35
  To determine the percentage of patients who achieve molecular remission and/or MRD negative remission by flow cytometry.
Events of special interest | 8 weeks post CAR NK, day +30 post HSCT
  To determine the rate of events of special interest including: Cytokine Release Syndrome, Immune Effector Cell Neurotoxicity Syndrome, Immune Effector Cell-Associated Hemophagocytic Lymphohistiocytosis-Like Syndrome, hepatic VOD, primary graft failure (in patients who undergo HSCT)
Neutrophil recovery | 1 year
  To evaluate the median time to neutrophil and platelet recovery

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Lamb, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided